CLINICAL TRIAL: NCT05226780
Title: A Prospective, Long-Term, Interventional, Active Extension Study to Evaluate the Safety and Tolerability of NBI-921352 as Adjunctive Therapy in Subjects With SCN8A Developmental and Epileptic Encephalopathy Syndrome (SCN8A-DEE)
Brief Title: Extension Study to Evaluate How Safe and Tolerable NBI-921352 is as an Adjunctive Therapy for Participants With SCN8A-DEE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-921352-DEE2013; 2021-004393-62 (EudraCT Number)
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: SCN8A Developmental and Epileptic Encephalopathy Syndrome
Keywords: Epilepsy; Sodium channel; voltage-gated; type VIII; alpha subunit (SCN8A); NaV1.6 inhibitor
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NBI-921352 (Experimental): NBI-921352 administered for up to 164 weeks.
  Interventions: Drug: NBI-921352

INTERVENTIONS:
Drug: NBI-921352 — Administered orally

SUMMARY:
Extension study to evaluate how safe and tolerable the drug NBI-921352 is when used as adjunctive therapy in participants with SCN8A developmental and epileptic encephalopathy syndrome (SCN8A-DEE).

ELIGIBILITY:
Key Inclusion Criteria:

For Participants Who Participated in NBI-921352-DEE2012:

* Written or oral pediatric assent from the participant and written informed consent from the participant's parent(s) or legal guardian(s) for pediatric participants and adult participants who are not capable of providing consent. Adult participant who are ≥18 years of age and capable of providing consent should sign an Informed Consent Form (ICF).
* Completed 16 weeks of treatment in Study NBI-921352-DEE2012.
* Continue to use a nocturnal alerting system or practice consistent with standards of care for the duration of the study.
* Have an adequate rescue medication regimen per the investigator's judgment in place for the duration of the study.

For Participants Who did not Participate in NBI-921352-DEE2012:

* Written or oral pediatric assent from the participant if deemed capable of providing assent and written informed consent from the participant's parent(s) or legal guardian(s) for pediatric participants and for adult participants who are not capable of providing consent. Adult participants who are capable of providing consent should sign an ICF.
* Be a male or female 2 to 21 years of age, inclusive.
* Have a diagnosis of SCN8A-DEE supported by both clinical and genetic findings.
* Have on average at least 1 countable motor seizure per week and not be seizure-free for more than 20 consecutive days.
* Being treated with at least 1 other antiseizure medication (ASM), but no more than 4 ASMs.
* Have failed to achieve seizure freedom with at least 2 ASMs.
* Have a body weight of at least 10 kilograms.

Key Exclusion Criteria

For Participants Who Participated in NBI-921352-DEE2012:

- Have developed any other disorder for which the treatment takes priority over treatment of SCN8A-DEE or is likely to interfere with study treatment or impair treatment compliance.

For Participants Who did not Participate in NBI-921352-DEE2012:

* Have symptoms that would be more consistent with another epilepsy disorder such as Dravet syndrome (for example, fever-induced episodes of status epilepticus, frequent myoclonic seizures, worsening on sodium channel blockers, absence seizures with generalized spike-and-wave electroencephalogram [EEG] as the sole seizure type).
* Currently receiving cannabinoids or medical marijuana except Epidiolex/Epidyolex, unless approved by the Sponsor.
* Currently taking systemic steroids (excluding inhaled medication for asthma treatments and intranasal steroids for allergies) such as adrenocorticotropin hormone, high-dose prednisolone for epileptic spasms. If participant has received these medications in the past, they must be off these medications for at least 3 months prior to the screening visit and these drugs may not be initiated during the duration of the study. Intermittent steroids to treat non-epilepsy-related diseases (such as allergies or dermatological conditions) are not exclusionary.
* Have a history of moderate or severe head trauma or other neurological disorders or systemic medical diseases that are, in the investigator's opinion, likely to affect nervous system functioning.
* Have a clinically significant medical condition or chronic disease, that in the opinion of the investigator would preclude the participant from participating in and completing the study or that could confound interpretation of study outcome.
* Have clinically significant abnormal vital signs at the screening visit, as determined by the investigator.
* Have one or more clinical laboratory test values outside the reference range, based on blood samples taken at the screening visit, that are of potential risk to the participants safety as determined by the investigator.
* Have, at the screening visit, an electrocardiogram (ECG) finding of a corrected QT interval using Fridericia's formula (QTcF) > 450 milliseconds (msec) or presence of any significant cardiac abnormality.

Ages: 2 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The participant incidence of serious treatment-emergent adverse events (TEAEs), TEAEs leading to discontinuation of study treatment, and fatal TEAEs | Day 1 to Week 168

SECONDARY OUTCOMES:
Percentage change from baseline in 28-day seizure frequency for countable motor seizures | Baseline, up to Week 162

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (4):
- United States (4):
  - UCSF Medical Center, San Francisco, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - University of Rochester, Rochester, New York
  - Cook Children's Medical Center, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No